CLINICAL TRIAL: NCT06174233
Title: "Contribution of Metagenomic Analysis of Faecal Microbiota Combined With Artificial Intelligence for the Prediction of Colorectal Cancer Risk; Study in Patients Scheduled for Colonoscopy".
Brief Title: The French Gut-colo
Status: Recruiting | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01941-44
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: Patients Aged 50-75 and Requiring Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Colorectal cancer (CRC) is the second most common type of cancer worldwide. The European Union recommends national CRC screening for people aged between 50 and 74. Generally, an immunological test called FIT (Fecal Immunochemical Test), based on the quantitative detection of human haemoglobin, is performed on a stool sample. If the haemoglobin level is above the recommended threshold, a colonoscopy is recommended to detect colorectal lesions. Recent studies have identified potential microbiota signatures associated with colon cancer. In this study, we will analyze the microbiota of a population aged 50 to 75 years undergoing colonoscopy as part of routine care in order to confirm the presence of microbiota signatures associated with the presence of adenomas, advanced adenomas and CRC.

DETAILED DESCRIPTION:
Many CRC risk factors, such as obesity, low physical activity, a diet low in fibre and high in fat and red meat, and chronic inflammation of the gastrointestinal tract, are known to interact with the intestinal microbiota. Recent studies have identified microbiota signatures associated with colon cancer. These CRC signatures could be used as a solid basis for future screening tests.

This study is an ancillary study of "Le French Gut" study (NCT05758961), a national contribution aiming to collect 100,000 faecal samples and associated nutritional and clinical data. Here, the aim is to identify microbiota profiles associated with the presence of adenomas, advanced adenomas and colorectal cancer (CRC), which would make it possible to recommend follow-up colonoscopies in a more targeted way than the current screening method. The study involves 2,500 patients aged between 50 and 75 who were due to undergo colonoscopy as part of their routine care. Patients recruited in this way will take part in the main "Le French Gut" study, will undergo a colonoscopy as part of their routine care and will complete 2 specific questionnaires relating to their personal and family history as well as their dietary habits in order to assess the risk factors for colorectal cancer as accurately as possible. The FIT test will be carried out as part of routine care with home sampling at the same time as stool sampling using the stool collection kit from the "French Gut" study (same stool sample).

Metagenomic fecal analysis will be coupled with a federated artificial intelligence tool incorporating data collected as part of the French Gut study and specific parameters describing the level of CRC risk. The diagnostic value of the signatures will be compared with that of the FIT test currently used for CRC screening.The ultimate aim is to develop more accurate, non-invasive ways of predicting CRC risk, based on a non-invasive fecal swab that can be taken at home.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 50 and 75
* Requiring colonoscopy
* Able to provide a faecal sample and to perform a FIT test prior to colonoscopy
* Without known inflammatory bowel disease (chronic inflammatory bowel disease (IBD), chronic ulcerative colitis (CUC) and Crohn's disease (CD))
* No medical condition that, in the opinion of the investigator, should preclude inclusion in the study
* Not having participated in any other clinical research study in which an investigational drug has been administered within 60 days prior to and including the date of informed consent or is likely to be administered during the period of colonoscopy
* Participation agreement signed electronically

Exclusion Criteria:

* Persons not living in France (declaratory);
* Persons subject to a protective measure, in particular guardianship or trusteeship, or unable to express their consent (declarative);
* Persons who have had a colectomy (declaratory);
* Person with a digestive stoma (declaration);
* Person who did not sign the consent form;
* Person who did not answer the entry questionnaire;
* Person who did not send a compliant stool sample;
* Antibiotics taken in the 3 months prior to inclusion (self-report);
* Person aged under 50 or over 75.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients aged between 50 and 75 scheduled for colonoscopy as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2028-06-25 (Estimated); Study Completion 2028-06-25 (Estimated)

PRIMARY OUTCOMES:
Measurement of true-negative, true-positive, false-negative and false-positive rates after colonoscopy, associated with the new test based on metagenomic analysis and clinical data. | up to 4 years

SECONDARY OUTCOMES:
Define and compare the true-negative, true-positive false-negative and false-positive rates after colonoscopy associated with the new test compared with those of the FIT test | up to 4 years
Compare the rates of true negatives, false-negative true positives and false-positives after colonoscopy associated with the new test with those of the FIT test: number of cases aggregated at 5 years, 10 years, 15 years and 20 years. | up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: ROBERT BENAMOUZIG, Pr, Principal Investigator — APHP
Locations (1):
- Hopital Avicenne, Centre de Recherche sur Volontaire, Bobigny, France

IPD SHARING:
Plan to Share IPD: No